CLINICAL TRIAL: NCT02236065
Title: A Pilot Study of Combination Therapy of Allogeneic Umbilical Cord Blood and Granulocyte-colony Stimulating Factor for Patients With Brain Injury or Neurodegenerative Disorders
Brief Title: Combination Therapy of Cord Blood and G-CSF for Patients With Brain Injury or Neurodegenerative Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MinYoung Kim, M.D. (Other)
Responsible Party: Sponsor-Investigator, MinYoung Kim, M.D., Professor, Bundang CHA Hospital
Organization: Bundang CHA Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCBnG-CSF
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Brain Injury; Cerebral Palsy; Amyotrophic Lateral Sclerosis; Parkinson's Disease
Keywords: Umbilical cord blood; Granulocyte-colony stimulating factor; Brain injury; Neurodegenerative disorder; Efficacy; Safety
MeSH Terms: conditions — Brain Injuries; Cerebral Palsy; Amyotrophic Lateral Sclerosis; Parkinson Disease; Neurodegenerative Diseases | interventions — Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- UCB + G-CSF (Experimental): UCB + G-CSF
  Interventions: Procedure: Umbilical cord blood therapy; Biological: Filgrastim

INTERVENTIONS:
Procedure: Umbilical cord blood therapy
Biological: Filgrastim

SUMMARY:
This open label trial is conducted to investigate the efficacy and safety of the combination therapy of allogeneic umbilical cord blood (UCB) and granulocyte-colony stimulating factor (G-CSF) for patients with brain injury or neurodegenerative disorders.

DETAILED DESCRIPTION:
Current treatments for brain injury or neurodegenerative disorders are palliative rather than curative. Preclinical and some clinical studies suggest that UCB and G-CSF can be used as restorative approach for such disorders.

ELIGIBILITY:
Inclusion Criteria: should be included one of the 4 disorders

* Brain injury: onset duration over 12 months, Age: 19 years or over
* Cerebral palsy: spastic, dyskinetic or ataxic, Age: 19 years or over
* Parkinson's disease: modified Hoehn and Yahr stage 2.5, 3, 4, Age: 30 to 75 years
* ALS: definite of possible ALS, progression during the past 6 months, Age: 19 to 65

Exclusion Criteria:

* Uncontrolled pulmonary, renal dysfunction at enrollment
* Uncontrolled seizure
* Malignant cancer
* Possibility of hypersensitivity to drugs used in this study
* Contraindication to the study intervention or assessment
* Pregnant or breast feeding women
* Non-compliance with the study visits specified in the protocol

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Changes in Berg Balance Scale | Baseline - 1 month - 3 months - 6 months
  Berg Balance Scale for brain injury and parkinson's disease (range: 0 to 56, Higher scores indicates better balance function.)
Changes in the Level of Disability | Baseline - 1 month - 3 months - 6 months
  FIM (Functional Independence Measure) for brain injury and cerebral palsy (range: 18 to 126, Higher scores indicate more independence in activities of daily living.)
Changes in Standardized Gross Motor Function | Baseline - 1 month - 3 months - 6 months
  GMFM (Gross Motor Function Measure) for cerebral palsy (range: 0 to 100, Higher scores indicate better gross motor function.)
Changes in Motor Performance | Baseline - 1 month - 3 months - 6 months
  GMPM (Gross Motor Performance Measure) for cerebral palsy (range: 0 to 100, Higher scores indicate better motor quality.)
Changes in ALSFRS-R | Baseline - 1 month - 3 months - 6 months
  ALSFRS-R (Amyotrophic Lateral Sclerosis Functional Rating Scale-revised) for ALS (range: 0 to 48, Higher scores indicate better physical function.)
Changes in UPDRS | Baseline - 1 month - 3 months - 6 months
  UPDRS (Unified Parkinson's Disease Rating Scale) for parkinson's disease (Part 1: mentation, behavior and mood; Part 2: activities of daily living; Part 3: motor examination; Part 4: complications of therapy; Part 5: Schwab and England activities of daily living scale)

SECONDARY OUTCOMES:
Changes in Brain MRI | Baseline - 6 months
  Analysis of Diffusion Tensor Image (DTI) for brain injury, cerebral palsy, ALS
Changes in Brain PET | Baseline - 6 months
  for parkinson's disease
Number of adverse events and participants with those adverse events | 6 months
  The numbers of adverse events and subjects with those serious adverse events within each group; A serious adverse event is any untoward medical occurrence that at any dose: results in death or is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or causes a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do, South Korea